CLINICAL TRIAL: NCT03517605
Title: Influence of a Rehabilitation Nursing Care Program on Quality of Life of Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Jorge Bravo, Principal Investigator, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evora
Record Dates: First submitted 2018-04-20; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Surgery Patients
Keywords: Cardiac Rehabilitation; Quality of Life; Rehabilitation Nursing
MeSH Terms: interventions — Exercise; Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: An exercise program was performed by the Specialist Nurses in Rehabilitation Nursing, comprising the combination of the various components of the exercise: aerobic and recovery/stretching. The program will start in the intensive care unit after the 24 hours post-surgery, and later, during hospitalization. The evaluations will be performed during hospitalization, in phase I of cardiac rehabilitation, and one-month post-discharge, in the Nursing visits of follow-up (phase II of cardiac rehabilitation). Clinical data (Blood Pressure, Heart Rate, Peripheral Oxygen Saturation) and Borg scale will be recorded in the initial, intermediate and final periods of each session. Capillary glycemia will be evaluated at the beginning of each session. Three sessions of exercises will be performed weekly with duration of 30 min to 60 min, divided in heating (10-25 min), aerobic exercise (10 min) and recovery (10-25min).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise for cardiac rehabilitation (Experimental): Three sessions of exercises will be performed weekly with duration of 30 min to 60 min, divided into heating, aerobic exercise and recovery.
  Interventions: Other: Exercise for cardiac rehabilitation

INTERVENTIONS:
Other: Exercise for cardiac rehabilitation — An exercise program was designed according to the American College of Sports Medicine and performed by the Specialist Nurses in Rehabilitation Nursing. Comprises aerobic and recovery/stretching. Started in the intensive care unit after the 24 hours post-surgery, and later, during hospitalization. Clinical data (Blood Pressure, Heart Rate, Peripheral Oxygen Saturation) and Borg scale will be recorded in the initial, intermediate and final periods of each session. Capillary glycemia will be evaluated at the beginning of each session. Three sessions of exercises will be performed weekly with duration of 30 min to 60 min, divided in heating (10-25 min), aerobic exercise (10 min) and recovery (10-25min). Possible symptoms will be controlled during exercise sessions.

SUMMARY:
Cardiac rehabilitation is fundamental in the treatment of patients undergoing cardiac surgery regarding the educational, physical exercise and quality of life dimensions. Considering the competences of Specialist Nurses in Rehabilitation Nursing and the current prevalence of risk factors associated with cardiovascular disease, it is essential to implement programs in this area.

This study aims to assess the impact of Specialist Nurses in Rehabilitation Nursing interventions on a cardiac rehabilitation program during hospitalization (phase I) and 1 month after cardiac surgery (phase II), in around 30 patients of both sexes, between 25 and 64 years old, and according to the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation, met the criteria for low or moderate risk, class B for participation and exercise supervision, absence of signs/symptoms after cardiac surgery, with a left ventricular ejection fraction greater than 40%. Supervised interventions were performed during hospitalization, pre- and post-cardiac surgery, and 1 month after hospital discharge. In phase II, a physical exercise program was fulfilled according to the norms of the American College of Sports Medicine, comprising 3 sessions of physical exercise per week lasting between 30 to 60 minutes, including heating, aerobic exercise, and recovery/stretching. Hemodynamic data (blood pressure, heart rate, peripheral oxygen saturation) and the Borg scale were recorded in the initial, intermediate and final periods of each session. The aerobic capacity was evaluated through the 6-Minute Walk Test and health-related quality of life using the Short Form Health Survey 36 (SF-36V2) questionnaire.

DETAILED DESCRIPTION:
Cardiac rehabilitation is fundamental in the treatment of patients undergoing cardiac surgery regarding the educational, physical exercise and quality of life dimensions. Considering the competences of Specialist Nurses in Rehabilitation Nursing and the current prevalence of risk factors associated with cardiovascular disease, it is essential to implement programs in this area.

Participants of both sexes will be included, between 25 and 64 years of age, meeting the criteria for low or moderate risk, class B for participation and exercise supervision, absence of signs/symptoms after cardiac surgery, with a left ventricular ejection fraction greater than 40%, according to the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation.

Inclusion criteria will consider patients with stable chronic heart failure (class I-III according to New York Heart Association), with dyslipidemia, controlled hypertension, without arrhythmias, without motor or psychic alterations, with previous acceptance of the informed consent of the intervention program. Participants will be excluded if present non-controlled arrhythmias, severe Chronic Obstructive Pulmonary Disease, uncontrolled high blood pressure, unstable angina, uncontrolled Diabetes Mellitus, decompensated coronary insufficiency, and pericarditis.

Supervised interventions will be provided during hospitalization, pre- and post-cardiac surgery, and 1 month after hospital discharge, considered phase I. In phase II, a physical exercise program will be performed, according to the norms of the American College of Sports Medicine, comprising 3 sessions of physical exercise per week lasting between 30 to 60 minutes, including heating, aerobic exercise and recovery/stretching. Hemodynamic data (blood pressure, heart rate, peripheral oxygen saturation) and the Borg scale will be recorded in the initial, intermediate and final periods of each session. The aerobic capacity will be evaluated through the 6-Minute Walk Test and health-related quality of life will be assessed through the Short Form Health Survey 36 (SF-36V2) questionnaire. No control will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients, between 25 to 64 years old, with stable chronic heart failure (class I-III according to NYCD); with dyslipidemia, controlled hypertension (AHT), without arrhythmias, without motor or psychic alterations, with previous acceptance of the informed consent of the intervention program.

Exclusion Criteria:

* Participants will be excluded if presents one or more of the following conditions: non-controlled arrhythmias, severe Chronic Obstructive Pulmonary Disease, uncontrolled high blood pressure, unstable angina, uncontrolled Diabetes Mellitus, decompensated coronary insufficiency, and pericarditis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in hemodynamic blood pressure in millimeters of mercury | 0,1 months
  Bruce treadmill protocol to assess hemodynamic blood pressure in response, in millimeters of mercury, after intervention in phase I and phase II of cardiac rehabilitation
Changes in hemodynamic heart rate in beats per minute | 0,1 months
  Bruce treadmill protocol to assess hemodynamic heart rate response, in beats per minute, after intervention in phase I and phase II of cardiac rehabilitation
Changes in hemodynamic peripheral oxygen saturation in percentage | 0,1 months
  Bruce treadmill protocol to assess hemodynamic peripheral oxygen saturation response, in percentage, after intervention in phase I and phase II of cardiac rehabilitation

SECONDARY OUTCOMES:
Changes in the perceived exertion between 6 to 20 points | 0,1 months
  Borg scale to assess perceived exertion, between 6 to 20 points, during intervention in phase I and phase II of cardiac rehabilitation.
Changes in the aerobic capacity in millilitres of oxygen per kilogram of body mass per minute | 0,1 months
  The 6-minute Walk Test to assess aerobic capacity, millilitres of oxygen per kilogram of body mass per minute, after intervention in phase I and phase II of cardiac rehabilitation
Changes in health-related quality of life questionnaire total score | 0,1 months
  The Short Form Health Survey 36 (SF-36V2) questionnaire total score to assess health-related quality of life after intervention in phase I and phase II of cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bravo, Ph.D., Principal Investigator — University of Évora; José Moreira, MSc, Principal Investigator — University of Évora
Locations (1):
- Universitry of Évora, Evora, Alentejo, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saji M, Katz MR, Ailawadi G, Welch TS, Fowler DE, Kennedy JLW, Bergin JD, Kuntjoro I, Dent JM, Ragosta M, Lim DS. 6-Minute walk test predicts prolonged hospitalization in patients undergoing transcatheter mitral valve repair by MitraClip. Catheter Cardiovasc Interv. 2018 Sep 1;92(3):566-573. doi: 10.1002/ccd.27600. Epub 2018 Apr 15. PMID 29656614
- [Background] Westerdahl E, Tenling A. Preoperative physical therapy reduces risk of postoperative atelectasis and pneumonia in people undergoing elective cardiac surgery. Evid Based Nurs. 2014 Jan;17(1):13-4. doi: 10.1136/eb-2012-101199. Epub 2013 Mar 6. No abstract available. PMID 23468240
- [Background] Mendis S, Davis S, Norrving B. Organizational update: the world health organization global status report on noncommunicable diseases 2014; one more landmark step in the combat against stroke and vascular disease. Stroke. 2015 May;46(5):e121-2. doi: 10.1161/STROKEAHA.115.008097. Epub 2015 Apr 14. No abstract available. PMID 25873596